CLINICAL TRIAL: NCT00781326
Title: Treatment of Depression Occurring in the Setting of Cerebrovascular Risk -- A Pilot Study
Brief Title: Effectiveness of Nimodipine Plus Antidepressant Medication in Treating Vascular Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Final cost of study medication was significantly greater than initial estimate,
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ellen Whyte, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23MH067710-01 (NIH); K23MH067710-01 (NIH); DATR AK-TNGP1
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Results first posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Depression
Keywords: Depressive Disorder, Major; Cerebrovascular Disorders; Risk Factors; Nimodipine
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Cerebrovascular Disorders | interventions — Nimodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label Antidepressant (Other): In Phase 1, all participants will be placed on antidepressant medication. In Phase 2, participants will continue with their antidepressant medication and also receive receive either nimodipine or placebo.
  Interventions: Drug: Nimodipine; Drug: Placebo

INTERVENTIONS:
Drug: Nimodipine — Nimodipine will be initiated at one, 30-mg tablet three times a day for 1 week, increased to 2 tablets three times a day for 1 week, and then increased to three tablets three times a day for the remaining 30 weeks of the study. Participants who cannot tolerate the maximum dose of 270 mg/day will be maintained at the highest tolerable dose.
  Other Names: Nimotop
Drug: Placebo — Placebo will be given in doses matching those of nimodipine.

SUMMARY:
This study will examine whether combined use of an antidepressant medication and the medication nimodipine reduces risk of depression relapse in patients with vascular depression.

DETAILED DESCRIPTION:
Depressed elderly patients often show signs of cerebrovascular disease, commonly known as a stroke. Some scientists theorize that having cerebrovascular disease may affect depression in older adults in one of three ways: by causing depression, by making it more likely that people who have been depressed have a relapse, or by maintaining certain depressive symptoms in those already depressed. The combination of depression and cerebrovascular disease in older adults is referred to as vascular depression and is associated with psychomotor slowing, functional impairment, and cognitive impairment. Additionally, the likelihood of improvement or remission is lower in vascular depression and is more difficult to treat over time.

Nimodipine (NIM) is FDA approved to reduce incidence and severity of problems with blood flow resulting from a particular type of stroke. In addition to improving blood flow in the brain following a stroke, NIM also protects neurons from injury or degeneration and has cognitive and functional benefits. These positive effects of NIM may make it useful for treatment of vascular depression. In a previous study of people with vascular depression, pairing NIM with the antidepressant fluoxetine showed greater improvements in depression treatment outcomes, higher likelihood of full remission, and less incidence of depression recurrence than using fluoxetine alone. This study will examine whether pairing NIM with other antidepressants will reduce recurrence of vascular depression.

Participation in this study will last 56 weeks and will be divided into two phases. In the first phase, participants will receive antidepressant medication without NIM. Participants will begin taking escitalopram but may be switched to duloxetine or have lorazepam added to their regimen, depending on individual treatment effectiveness and side effects. The first phase will last between 6 and 24 weeks, ending when the individual participant either responds to medication or experiences 24 weeks of nonresponse. During the first phase, participants will attend weekly study visits, during which researchers will assess medication effectiveness and monitor side effects.

At the beginning of the second phase, participants will be randomly assigned to receive either NIM or a placebo in addition to continuing with the antidepressant medication already helping them. Participants will take NIM or the placebo for 8 months, undergoing weekly study visits for the first month and monthly study visits for the last 7 months. During these visits, researchers will monitor the participants' health and reactions to their medications. After 4, 16, and 32 weeks, an EKG test will be performed, and after 16 and 32 weeks, cognitive and physical tests will be performed again. After the 8 months, participants will attend three weekly study visits while their use of medication is lowered and then ended.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00177424

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-IV (Diagnostic and Statistical Manual) diagnosis of major depression
* Score greater than 15 on the 24-item Hamilton Depression Rating Scale (HDRS24)
* Significant cerebrovascular disease risk factors, as defined by the presence of more than three of the following:

  1. Arterial hypertension, defined by a systolic blood pressure higher than 140 mm Hg or a diastolic blood pressure higher than 90 mm Hg, or by both a self-reported hypertension diagnosis and use of antihypertensive medication
  2. Diabetes mellitus, defined by a fasting blood glucose level higher than 126 mg/dl or treatment with hypoglycemic agents or insulin in the year before study entry
  3. Obesity, defined by a current body mass index (BMI) greater than 30
  4. Hyperlipidemia, defined by either a confirmed prior diagnosis or a current fasting cholesterol level higher than 200 mg/dl
  5. Current smoker
* Able to swallow oral medication
* Identification of a family member or friend willing and able to participate as a source of corroborating information
* Able to speak English
* A hearing capacity adequate to respond to a raised conversational voice

Exclusion Criteria:

* Current diagnosis of major depression with psychosis, schizophrenia, bipolar disorder, schizophreniform disorder, schizoaffective disorder, schizotypal disorder, or obsessive compulsive disorder
* Meets DSM-IV criteria for dementia or has a score of 17 or lower on the Mini Mental State Examination
* Met DSM-IV criteria for drug or alcohol dependence within the past 6 months
* Not responsive to therapeutic trials of either escitalopram or duloxetine for the current major depressive episode
* Acute, severe, or unstable medical disorder likely to interfere with treatment, such as untreated thyroid disorder
* History of epilepsy
* Clinically reported stroke within the past year
* First-degree heart block, determined after correcting for age
* Symptomatic hypotension or symptomatic orthostatic hypotension
* History of nontolerance or allergy to both escitalopram and duloxetine therapy, including history of selective serotonin reuptake inhibitor (SSRI)-related syndrome of inappropriate anti-diuretic hormone secretion (SIADH)
* Significant allergy to NIM or other ingredients contained in the study medication
* Taken monoamine oxidase inhibitors (MAOIs) within the 2 weeks prior to the first administration of double-blind study medication
* Requires treatment with amiodarone, protease inhibitors, dalfopristin or quinupristin, valproic acid, triazole antifungal agents (e.g., itraconazole), reserpine, methyldopa, guanethidine, or clonidine during the course of the study
* May require drugs known to interact with NIM during the course of the study
* Refusal to allow the research team to contact participant's primary medical provider
* Planning to become pregnant during the course of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M. Whyte, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Taragano FE, Bagnatti P, Allegri RF. A double-blind, randomized clinical trial to assess the augmentation with nimodipine of antidepressant therapy in the treatment of "vascular depression". Int Psychogeriatr. 2005 Sep;17(3):487-98. doi: 10.1017/s1041610205001493. PMID 16252380
- [Background] Alexopoulos GS, Meyers BS, Young RC, Campbell S, Silbersweig D, Charlson M. 'Vascular depression' hypothesis. Arch Gen Psychiatry. 1997 Oct;54(10):915-22. doi: 10.1001/archpsyc.1997.01830220033006. PMID 9337771
- [Background] Coffey CE, Figiel GS, Djang WT, Weiner RD. Subcortical hyperintensity on magnetic resonance imaging: a comparison of normal and depressed elderly subjects. Am J Psychiatry. 1990 Feb;147(2):187-9. doi: 10.1176/ajp.147.2.187. PMID 2301657
- [Background] Figiel GS, Krishnan KR, Doraiswamy PM, Rao VP, Nemeroff CB, Boyko OB. Subcortical hyperintensities on brain magnetic resonance imaging: a comparison between late age onset and early onset elderly depressed subjects. Neurobiol Aging. 1991 May-Jun;12(3):245-7. doi: 10.1016/0197-4580(91)90104-r. PMID 1876230
- [Background] Hickie I, Scott E, Mitchell P, Wilhelm K, Austin MP, Bennett B. Subcortical hyperintensities on magnetic resonance imaging: clinical correlates and prognostic significance in patients with severe depression. Biol Psychiatry. 1995 Feb 1;37(3):151-60. doi: 10.1016/0006-3223(94)00174-2. PMID 7727623
- [Background] Simpson SW, Jackson A, Baldwin RC, Burns A. 1997 IPA/Bayer Research Awards in Psychogeriatrics. Subcortical hyperintensities in late-life depression: acute response to treatment and neuropsychological impairment. Int Psychogeriatr. 1997 Sep;9(3):257-75. doi: 10.1017/s1041610297004432. PMID 9513027
- [Background] Simpson S, Baldwin RC, Jackson A, Burns A, Thomas P. Is the clinical expression of late-life depression influenced by brain changes? MRI subcortical neuroanatomical correlates of depressive symptoms. Int Psychogeriatr. 2000 Dec;12(4):425-34. doi: 10.1017/s1041610200006542. PMID 11263709

RESULTS

PARTICIPANT FLOW:
Period: Phase I
Arm/Group | Open Label Antidepressant
Started | 6 (Nine subjects consented; 3 did not meet eligibility criteria. 6 started antidepressant treatment.)
Completed | 2
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2
Period: Phase 2
Arm/Group | Open Label Antidepressant
Started | 0 (Study terminated prior to enrollment into Phase II)
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Antidepressant
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Hamilton Depression Rating Scale (24 item) [Mean (Standard Deviation); unit: units on a scale] — Hamilton Depression Rating Scale (24 item) measures symptoms of major depression. We report total score which is the sum of all items. Total score range is 0 to 76 with higher scores indicating more severe depression.
  units on a scale | 20.5 (2.4)
Cumulative Illness Rating Scale (Geriatric) total [Mean (Standard Deviation); unit: units on a scale] — Cumulative Illness Rating Scale (Geriatric Version) is a measure of medical illness burden across 14 body systems. For the purposes of this study, we do not include the "psychiatric body system". Within each body system, the burden of medical illness is scored 0 - 4. The total score reported here is the sum of medical burden scores across 13 body systems. Total score range is 0 to 52 with higher scores indicating greater overall burden of medical illness.
  units on a scale | 8.3 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (24 Item) [Phase I Primary Outcome]
Description: Hamilton Depression Rating Scale (24 item) measures symptoms of major depression. We report total score which is the sum of all items. Total score range is 0 to 76 with higher scores indicating more severe depression. We reports scores at end of Phase I for subjects completing the phase.
Time Frame: End of Phase I (at 24 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Antidepressant
Number analyzed (Participants) | 2
units on a scale | 9.5 (0.7)

ADVERSE EVENTS:
Time Frame: Phase I (at or before 24 weeks)
Arm/Group | Open Label Antidepressant
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Antidepressant (N=6)
Mania (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated for administrative reasons at the end of Phase I (open label antidepressant treatment). No subjects entered Phase II (Nimodipine vs Placebo).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No